CLINICAL TRIAL: NCT01273688
Title: Eccentric Training With Our Without Elbow Brace for Epicondylitis - a Randomized Clinical Trial
Brief Title: Eccentric Training With or Without Elbow Brace for Epicondylitis
Acronym: EpiFlex
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Hannover Medical School, Karsten Knobloch, FACS, MD, PhD, Hannover Medical School, Plastic, Hand and Reconstructive Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EpiFlex
Record Dates: First submitted 2011-01-03; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Epicondylitis; Tendinopathy; Pain
Keywords: pain; elbow; tendinopathy
MeSH Terms: conditions — Tendinopathy; Pain | interventions — Braces; Orthotic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eccentric training only (Active Comparator): Eccentric training only active control group (Flex-Bar)
  Interventions: Behavioral: Eccentric training (Flex-Bar)
- Eccentric training and elbow brace (Experimental): Combined eccentric training (Flex-Bar) and elbow brace (Epi-Hit)
  Interventions: Behavioral: Eccentric training (Flex-Bar); Device: EpiHit elbow brace

INTERVENTIONS:
Behavioral: Eccentric training (Flex-Bar) — 6x15 repetitions of supination and pronation daily over 12 weeks
Device: EpiHit elbow brace — daily wearing of the EpiHit elbow brace
  Other Names: brace; orthosis; strap
  Arms: Eccentric training and elbow brace

SUMMARY:
Lateral epicondylitis is a painful overuse condition also described as lateral elbow tendinopathy. As at the Achilles tendon or the patella tendon, lateral elbow tendinopathy has striking clinically and histologically similarities. As such, neovascularisation closely related to pain-mediating fibers are encountered. Eccentric painful exercise is of clinical use in Achilles and patella tendinopathy. We sought to evaluate the clinical effect of a painful eccentric training (supination and pronation) with or without a orthopedic elbow brace in lateral epicondylitis.

DETAILED DESCRIPTION:
Two study arms are planned with both groups performed a home-based eccentric training using a Thera-Band Flex-Bar device. Supination and pronation are performed with each position on hold for 2s with 15 repetitions. This is repeated in three sets of 15 repetitions each twice daily. In other words, 6x15 repetitions of supination and pronation per day are suggested in the eccentric training using the Thera-Band Flex-Bar.

The combination group performs the same eccentric training. In addition, patients wear a orthopedic elbow brace (Epi-Hit) in order to overcome the elbow pain.

This is a clinical trial, thus pain reduction on a visual analogue scale is the primary outcome parameter. Evaluation will be performed after 12 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* lateral elbow tendinopathy
* 18-80 years informed consent

Exclusion Criteria:

* no elbow tendinopathy <18 or > 80 years no informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Pain on visual analogue scale (VAS 0-10) | 12 weeks
  Pain on VAS (0=no pain, 10=worst pain)

SECONDARY OUTCOMES:
Grip strength (JAMAR) | 12 weeks
  Grip strength (JAMAR, kg) in two elbow positions: 0° flexion and 90° flexion
Elbow microcirculation | 12 weeks
  Oxygen-to-see combined Laser-Doppler flowmetry and spektrophotometry system non-invasively analyzing three parameters: tissue oxygen saturation, capillary blood flow, postcapillary venous filling pressure
DASH Score [0-100] | 12 weeks
  DASH score [0=no impairment of daily activities, 100= severe impairment) before and 12 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Knobloch, FACS, MD, PhD, Principal Investigator — Hannover Medical School, Germany
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Background] Garg R, Adamson GJ, Dawson PA, Shankwiler JA, Pink MM. A prospective randomized study comparing a forearm strap brace versus a wrist splint for the treatment of lateral epicondylitis. J Shoulder Elbow Surg. 2010 Jun;19(4):508-12. doi: 10.1016/j.jse.2009.12.015. Epub 2010 Apr 2. PMID 20363158
- [Background] Knobloch K, Gohritz A. Dr Runge: a German pioneer in sclerosing therapy in epicondylitis in 1873. Br J Sports Med. 2010 Nov 16. doi: 10.1136/bjsm.2008.051326. Online ahead of print. No abstract available. PMID 21081643
- [Background] Knobloch K. [Non-operative therapy in lateral epicondylitis]. MMW Fortschr Med. 2009 Feb 19;151(8):28-30. No abstract available. German. PMID 19432271
- [Background] Knobloch K. Re: Radiofrequency microtenotomy: a promising method for treatment of recalcitrant lateral epicondylitis. Am J Sports Med. 2008 Nov;36(11):e2-3; author reply e3. doi: 10.1177/0363546508325661. No abstract available. PMID 18978181
- [Background] Knobloch K. Lateral elbow tendinopathy. Am J Sports Med. 2010 Nov;38(11):NP3; author reply NP3-4. doi: 10.1177/0363546510383492. No abstract available. PMID 20971969
- [Background] Knobloch K, Spies M, Busch KH, Vogt PM. Sclerosing therapy and eccentric training in flexor carpi radialis tendinopathy in a tennis player. Br J Sports Med. 2007 Dec;41(12):920-1. doi: 10.1136/bjsm.2007.036558. Epub 2007 May 11. PMID 17496066
- [Background] Knobloch K, Kramer R, Redeker J, Spies M, Vogt PM. [Scaphoid fracture in motocross riders]. Sportverletz Sportschaden. 2009 Dec;23(4):217-20. doi: 10.1055/s-0028-1109927. Epub 2009 Dec 15. German. PMID 20108186
- [Background] Knobloch K, Schreibmueller L, Kraemer R, Jagodzinski M, Vogt PM, Redeker J. Gender and eccentric training in Achilles mid-portion tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2010 May;18(5):648-55. doi: 10.1007/s00167-009-1006-7. Epub 2009 Dec 9. PMID 19997901
- [Background] Kramer R, Lorenzen J, Vogt PM, Knobloch K. [Systematic review about eccentric training in chronic achilles tendinopathy]. Sportverletz Sportschaden. 2010 Dec;24(4):204-11. doi: 10.1055/s-0029-1245820. Epub 2010 Dec 14. German. PMID 21157656
- [Background] Lorenzen J, Kramer R, Vogt PM, Knobloch K. [Systematic review about eccentric training in chronic patella tendinopathy]. Sportverletz Sportschaden. 2010 Dec;24(4):198-203. doi: 10.1055/s-0029-1245818. Epub 2010 Dec 14. German. PMID 21157655
- [Background] Knobloch K, Hufner T. [Conservative treatment of Achilles tendinopathy]. Unfallchirurg. 2010 Sep;113(9):705-11. doi: 10.1007/s00113-010-1808-6. German. PMID 20725821
- [Background] Knobloch K. Eccentric training and the science behind. Med Sci Sports Exerc. 2009 Jan;41(1):251; author reply 252. doi: 10.1249/MSS.0b013e31818cae4b. No abstract available. PMID 19106784
- [Background] Knobloch K, Gohritz A, Spies M, Vogt PM. Neovascularisation in de Quervain's disease of the wrist: novel combined therapy using sclerosing therapy with polidocanol and eccentric training of the forearms and wrists-a pilot report. Knee Surg Sports Traumatol Arthrosc. 2008 Aug;16(8):803-5. doi: 10.1007/s00167-008-0555-5. Epub 2008 May 31. PMID 18516593